CLINICAL TRIAL: NCT03432936
Title: Prospective Use of Philips iSuite for Interventional Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, David A. Woodrum, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-007674
Record Dates: First submitted 2018-01-02; First posted 2018-02-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MRI guided procedure software evaluation (Experimental): Evaluate the workflow and effectiveness of the Philips Interventional iSuite software during biopsies and/or ablations versus standard MR imaging in aiding needle placement.
  Interventions: Device: MRI guided procedure software evaluation

INTERVENTIONS:
Device: MRI guided procedure software evaluation — MRI guided ablation/biopsy using standard MR imaging along with Philips Interventional iSuite software tools.

SUMMARY:
This research study is being done to look at new MRI imaging guidance software, Philips Interventional iSuite software, to see if using will improve the physician's ability to quickly place and guide needle tip position for biopsies and ablations.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate Philips Interventional iSuite software used for MRI guided procedures in the MRI suite. The real-time MRI Imaging software will be used during an MRI procedure to take continuous pictures.

The Philips Interventional iSuite software package has not received FDA 510(k) clearance. The Investigator will be evaluating and publishing on the use of this software as a clinical aid in performing interventional procedures within the MR suite. The primary evaluation will be weighted toward enhanced facilitation of ablation procedures. However, the software will not replace standard MR imaging for final confirmation of needle tip position and ablation margins.

ELIGIBILITY:
Inclusion criteria:

* Patients already scheduled for a percutaneous MR guided procedure

Exclusion criteria:

* Pregnant Women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Needle placement efficiency into target lesion | Will assess for 3 years with interval assessment each year
  Needle placement efficiency record time to final needle position, and compare overall similarity of use with current CT guided intervention during the interventional procedure in order to determine how the iSuite may facilitate intervention with the MRI environment. Each operator will fill out a short questionnaire after each intervention.

SECONDARY OUTCOMES:
Software ease of use in targeting lesion for treatment | Will assess for 3 years with interval assessment each year
  Evaluate the ease of use of the software for needle placement

CONTACTS AND LOCATIONS:
Overall Officials: David A Woodrum, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials